CLINICAL TRIAL: NCT03302039
Title: Three Protocols for Phenylephrine Administration for Prophylaxis Against Post-spinal Hypotension During Cesarean Delivery
Brief Title: Three Protocols for Phenylephrine Administration in Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: N-71-2017
Record Dates: First submitted 2017-10-01; First posted 2017-10-04 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Cesarean Section Complications; Spinal Anesthesia
MeSH Terms: interventions — Phenylephrine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single shot (Experimental): Spinal anesthesia will be performed using intrathecal bupivacaine. Then, a single shot phenylephrine (1.5 ug/Kg) will be administered.
  Interventions: Drug: Single shot phenylephrine; Drug: Bupivacaine
- Fixed infusion (Active Comparator): Spinal anesthesia will be performed using intrathecal bupivacaine. Then, fixed infusion phenylephrine will be administered at a dose of (0.75 mcg/Kg/min). the infusion will stop if reactive hypertension occurred.
  Interventions: Drug: Fixed infusion phenylephrine.; Drug: Bupivacaine
- Variable infusion (Active Comparator): Spinal anesthesia will be performed using intrathecal bupivacaine. Then, variable infusion phenylephrine will be administered at a starting dose of (0.75 mcg/Kg/min). the infusion will be titrated according to blood pressure.
  Interventions: Drug: Variable infusion phenylephrine.; Drug: Bupivacaine

INTERVENTIONS:
Drug: Single shot phenylephrine — A single shot of phenylephrine (1.5 mcg/Kg) will be administrated intravenously.
  Other Names: Phenylephrine
  Arms: Single shot
Drug: Fixed infusion phenylephrine. — Fixed infusion of phenylephrine will be administrated at a rate of 0.75 mcg/Kg/min
  Other Names: Phenylephrine
  Arms: Fixed infusion
Drug: Variable infusion phenylephrine. — Variable infusion of phenylephrine will be administrated at a starting rate of 0.75 mcg/Kg/min.
  Other Names: Phenylephrine
  Arms: Variable infusion
Drug: Bupivacaine — Bupivacaine will be administrated in the subarachnoid space for spinal anesthesia.
  Other Names: Marcaine

SUMMARY:
The investigators will compare variable infusion of phenylephrine (at a starting rate of 0.75 mcg/Kg/min) with fixed rate (0.75 mcg/Kg/min which will stop of reactive hypertension occurred) and single shot (1.5 mcg/Kg) phenylephrine.

DETAILED DESCRIPTION:
Maternal hypotension is a common complication after spinal anesthesia for cesarean delivery (CD). Phenylephrine (PE) is the most popular vasopressor for prevention of post-spinal hypotension (PSH) during CD; however, the most appropriate protocol for PE administration is still unknown. The most common PE protocols used for prophylaxis against PSH are: single shot, fixed infusion, and variable infusion. A recent study reported that a dose of 1.5 mcg/Kg is the most suitable single-shot dose for prophylaxis. Another randomized controlled trial compared four doses of PE infusion and reported that 25 mcg/Kg/min and 50 mcg/Kg/min doses were the best doses for fixed infusion with accepted incidence of both PSH as well as reactive hypertension. Using variable infusion rate of PE had been recently introduced in another study with a starting dose of 0.75 mcg/Kg/min. The variable rate infusion showed very good results regarding PSH. In this study, the investigators will compare variable infusion of PE (at a starting rate of 0.75 mcg/Kg/min) with fixed rate (0.75 mcg/Kg/min which will stop if reactive hypertension occurred) and single shot protocol (1.5 mcg/Kg).

ELIGIBILITY:
Inclusion Criteria:

* Full term
* Pregnant women
* Scheduled for cesarean delivery

Exclusion Criteria:

* Pre-eclampsia
* Eclampsia
* Hemorrhage
* Cardiac dysfunction
* Baseline low heart rate (below 60 bpm)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 217 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Post-spinal anesthesia hypotension | 30 minutes after spinal anesthesia
  Defined as percentage of patients with decreased systolic blood pressure less than 80% of the baseline reading during the period from intrathecal injection to delivery of the fetus

SECONDARY OUTCOMES:
Incidence of severe Post-spinal anesthesia hypotension | 30 minutes after spinal anesthesia
  Defined as percentage of patients with decreased systolic blood pressure less than 60% of the baseline reading during the period from intrathecal injection to delivery of the fetus.
Incidence of reactive hypertension | 2 hours after spinal anesthesia
  Defined as percentage of patients with increased systolic blood pressure more than 80% of the baseline reading during the period from intrathecal injection to delivery of the fetus.
Systolic blood pressure | 2 hours after spinal anesthesia
  Systolic blood pressure measured in mmHg
Diastolic blood pressure | 2 hours after spinal anesthesia
  Diastolic blood pressure measured in mmHg
Heart rate | 2 hours after spinal anesthesia
  number of heart beats per minute
APGAR score | 10 minutes after delivery
  APGAR score of the fetus
umbilical arterial PH | 10 minutes after delivery
  the PH in umbilical arterial blood
umbilical arterial Pco2 | 10 minutes after delivery
  umbilical arterial Pco2 measured in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mukhtar, Professor, Study Director — Head of research committee section in anesthesia department
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided